CLINICAL TRIAL: NCT05143957
Title: A Phase 2a, Randomized, Open-Label Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 702843 Administered to Patients With Phlebotomy Dependent Polycythemia Vera (PD-PV)
Brief Title: A Study to Evaluate Sapablursen (Formerly ISIS 702843, IONIS-TMPRSS6-LRx) in Patients With Polycythemia Vera
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 702843-CS4; 2021-003704-40 (EudraCT Number)
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Phlebotomy Dependent Polycythemia Vera
Keywords: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sapablursen Dose Level 1 (Experimental): Sapablursen will be administered by SC injection every 4 weeks.
  Interventions: Drug: sapablursen
- Sapablursen Dose Level 2 (Experimental): Sapablursen will be administered by SC injection every 4 weeks
  Interventions: Drug: sapablursen

INTERVENTIONS:
Drug: sapablursen — Sapablursen will be administered by SC injection.
  Other Names: ISIS 702843; IONIS-TMPRSS6-LRx

SUMMARY:
The main purpose of this study is to evaluate the efficacy of sapablursen in reducing the frequency of phlebotomy and in improving quality of life assessments in participants with polycythemia vera.

DETAILED DESCRIPTION:
This is a Phase 2a, multi-center, randomized, open-label study of sapablursen in up to 40 participants with PD-PV. The study consists of 4 periods: 1) Screening Period: up to 7 weeks; 2) Treatment Period: 37 weeks 3) Treatment Extension Period: 36 weeks; 4) Post-treatment Period: 13 weeks.

In the Treatment Period, study drug is given by subcutaneous (under the skin) injection(s). There will be a total of 9 doses given over about 8 months.

In the Treatment Extension Period, there will be a total of 9 doses given over about 8 months.

Participants will be assigned to receive one of 2 Dosing Levels - a higher or a lower level, with an equal chance of being assigned to either Dosing Level. All participants will receive study drug; there is no placebo.

This study was extended to allow participants to receive sapablursen for an additional 36 weeks following the initial 37-week treatment period.

ELIGIBILITY:
Inclusion Criteria

1. Meet modified World Health Organization (WHO) 2016 diagnostic criteria for polycythemia vera (PV) at the time of clinical diagnosis
2. Participant must be phlebotomy dependent.
3. Participants do not need to be on cytoreductive therapy and do not need to have been previously treated with cytoreductive therapy. If the patient was previously on cytoreductive therapy it must have been discontinued at least 3 months prior to Screening, with all associated AEs resolved. If the patient is currently on cytoreductive therapy they must be on a stable dose of hydroxyurea, recombinant or PEGylated interferon, or ruxolitinib for at least 3 months prior to Screening.

Exclusion Criteria

1. Meets criteria for post-polycythemia vera myelofibrosis (PPV-MF) as defined by the International Working Group- Myeloproliferative Neoplasms Research and Treatment (IWG-MRT)
2. Moderate to severe splenic pain or spleen-related organ obstruction
3. Active or chronic bleeding within 1 month of Screening, significant concurrent/recent coagulopathy, history of immune thrombocytopenic purpura (ITP)
4. Known primary or secondary immunodeficiency
5. Active infection with human immunodeficiency virus (HIV), hepatitis C, or hepatitis B.
6. Active infection requiring systemic antiviral or antimicrobial therapy or active novel coronavirus disease (Covid-19) infection
7. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or non-metastatic prostate cancer that has been successfully treated
8. Surgery requiring general anesthesia within 1 month prior to Screening

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the frequency of phlebotomy comparing Baseline with the last 20 weeks of the 37 week Treatment Period | Week 17 to Week 37

SECONDARY OUTCOMES:
Proportion of patients achieving a reduction in the frequency of phlebotomy by ≥ 30%, ≥ 50%, ≥ 75% and ≥ 90% comparing Baseline with the last 20 weeks of the 37-week Treatment Period | Week 17 to Week 37
Change in the Myeloproliferative Neoplasm Symptom Assessment Form-Total Symptom Score (MPN-SAF-TSS) From Baseline to Week 37 | Baseline up to Week 37

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - O'Neal Comprehensive Cancer Center University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Border Medical Oncology Research Unit, Albury
- McGill University Health Centre, Montreal, Quebec, Canada
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie, Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
  - Wojewódzki Szpital Specjalistyczny Sp. z o.o., Słupsk
  - MICS Centrum Medyczne Toruń, Torun
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/